CLINICAL TRIAL: NCT05686863
Title: Sedative Effect and Safety of Remiazolam Combined With Low-dose Esketamine in Painless Bidirectional Endoscopy in Children
Brief Title: Remiazolam Combined With Esketamine in Painless Bidirectional Endoscopy in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tongji Hospital (Other)
Responsible Party: Principal Investigator, aijun xu, Dr. aijun Xu, Tongji Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RECES
Record Dates: First submitted 2023-01-07; First posted 2023-01-17 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Drug Effect
Keywords: remiazolam; esketamine; bidirectional endoscopy; children
MeSH Terms: interventions — remimazolam; Esketamine; Propofol; Remifentanil

STUDY DESIGN:
Intervention Model Description: Prospective, randomized controlled study
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Since propofol is white uniform emulsion, and ramazolam is colorless, clear and transparent liquid, anesthesiologists and surgeons may see the color of the study drug during operation, so this study is a single blind clinical study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P group (Active Comparator): induction: Propofol 3 mg/kg+Esketamine 0.25 mg/kg intravenously, mantainance: propofol 5-10 mg/kg/h+remifentanil 0.5-1 μg/kg/h continuous pumping
  Interventions: Drug: Esketamine; Drug: Propofol; Drug: remifentanil
- R group (Experimental): induction: Remimazolam 0.3 mg/kg+Esketamine 0.25 mg/kg intravenously, mantainance: Remimazolam 1-3 mg/kg/h+remifentanil 0.5-1 μg/kg/h continuous pumping
  Interventions: Drug: Remimazolam; Drug: Esketamine; Drug: remifentanil

INTERVENTIONS:
Drug: Remimazolam — Remazolam for sedation in children undergoing bidirectional endoscopy
  Other Names: Rema
  Arms: R group
Drug: Esketamine — Esketamine
  Other Names: Esket
Drug: Propofol — Propofol
  Other Names: Prop
  Arms: P group
Drug: remifentanil — remifentanil
  Other Names: remifen

SUMMARY:
To observe the sedative effect and safety of remiazolam combined with small dose of esketamine in painless bidirectional endoscopy in children, and to provide a more reasonable and safe sedative and analgesic regimen for children's gastrointestinal endoscopy.

DETAILED DESCRIPTION:
It is planned to observe the painless two-way endoscopic examination of children in Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology from November 2022 to May 2023.To observe the sedative effect and safety of remiazolam combined with small dose of esketamine in painless bidirectional endoscopy in children, and to provide a more reasonable and safe sedative and analgesic regimen for children's gastrointestinal endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-17;
* ASA Class I-II;
* Sign the informed consent form.

Exclusion Criteria:

* Patients with high risk of stomach satiety and reflux aspiration;
* Patients allergic to the study drug;
* Obesity or severe malnutrition;
* Those who have taken sedative, analgesic or antidepressant drugs within 24 hours;
* Hypertension without treatment;
* Abnormal liver and kidney function (index ≥ 2 times the upper limit of normal reference range);
* Other congenital diseases or acute and chronic diseases that affect the observation of curative effect;
* Participate in other clinical studies within 4 weeks.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 106 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2023-07-07 (Actual); Study Completion 2023-07-07 (Actual)

PRIMARY OUTCOMES:
Sedation success rate | Procedure (From the beginning of anesthesia to the end of examination)
  Improved observer alertness and sedation score, MOAA/S

CONTACTS AND LOCATIONS:
Overall Officials: Hong Liu, Dr, Study Director — Tongji Hospital
Locations (1):
- Tongji Hospital, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No
Research data can be requested from the main researchers via email

REFERENCES:
- [Derived] Chu T, Zhou S, Wan Y, Liu Q, Xin Y, Tian Z, Yan T, Xu A. Comparison of remimazolam and propofol combined with low dose esketamine for pediatric same-day painless bidirectional endoscopy: a randomized, controlled clinical trial. Front Pharmacol. 2024 Feb 5;15:1298409. doi: 10.3389/fphar.2024.1298409. eCollection 2024. PMID 38375038